CLINICAL TRIAL: NCT04733378
Title: Impact of Surgical Timing on the Neurodevelopmental Prognosis of Newborns With Complex Congenital Heart Disease
Acronym: CINC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-44; 2020-A00369-30 (Other: ANSM)
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Complex Congenital Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peri-operative neurological monitoring (Experimental)
  Interventions: Procedure: Peri-operative neurological monitoring

INTERVENTIONS:
Procedure: Peri-operative neurological monitoring — Pre- and post-operative cerebral MRI, standardized neurological examinations at 4, 12, 24 months and neuropsychological evaluation with a Bayley III test (Bayley Scale of Infant and Toddler Development, Third Edition) at 24 months.

SUMMARY:
We propose a prospective observational study whose main objective will be to determine whether there is an association between age at surgery (days of life) and neurodevelopmental outcome in patients with CCHD. Secondly, we will study the relationship between age at surgery and (i) the incidence of WMI observed on pre- and post-operative cerebral MRI (ii) post-operative morbidity as defined by the occurrence of post-operative complications (haemodynamic, infectious, neurological, surgical) and (iii) the length of hospital stay.

DETAILED DESCRIPTION:
Congenital heart disease is the most frequent congenital malformation and concerns 9 newborns per 1000 live births, i.e. nearly 1% of births. Half of these children present a complex form of congenital heart disease requiring surgery during the first months of life. More than one child in two will present a neurodevelopmental disorder resulting from brain damage beginning in utero and continuing in the post-natal period. In the newborn with complex congenital heart disease (CCHD), cerebral immaturity is synonymous with vulnerability, leading in half of the cases to the perioperative occurrence of hypoxic-ischemic cerebral lesions, most of which affect the white matter. These white matter injuries (WMI) are a prognostic factor for motor, cognitive, language and behavioural disorders that induce psycho-social difficulties in adulthood, altering the quality of life of patients. In newborns with CCHD (Transposition of Great Arteries or Left Ventricular Hypoplasia) operated on later in the neonatal period, both the incidence of perioperative BSL and post-operative morbidity are increased.

Earlier surgery may therefore be a neuroprotective strategy leading to a reduction in perioperative WMI, postoperative morbidity and a better neurodevelopmental prognosis in infants with CCHD.

The investigators propose a prospective observational study whose main objective will be to determine whether there is an association between age at surgery (days of life) and neurodevelopmental outcome in patients with CCHD. Secondly, the investigators planned to study the relationship between age at surgery and (i) the incidence of WMI observed on pre- and post-operative cerebral MRI (ii) post-operative morbidity as defined by the occurrence of post-operative complications (haemodynamic, infectious, neurological, surgical) and (iii) the length of hospital stay.

Recruitment will be performed in a prospective cohort (n=50) of neonates with CCHD requiring surgery during the first 2 months of life and benefiting from pre- and post-operative cerebral MRI, standardized neurological examinations at 4, 12, 24 months and neuropsychological evaluation with a Bayley III test at 24 months.

ELIGIBILITY:
Inclusion criteria

* Patients aged 2 months or less with complex congenital heart disease (CCHD) requiring surgery with cardiac circulation during their first 2 months of life
* Eligible heart diseases: Transposition of the Large Vessels (TGV), hypoplasia of the left ventricle, right ventricle with double outlet type Fallot or TGV, obstruction of the aortic arch, truncus arteriosus, atrioventricular duct, pulmonary atresia with or without communication inter ventricular.
* Informed consent signed by both parents
* Patient affiliated to health social security

Non-inclusion criteria:

* patients with a birth weight less than 2 kilograms and / or a gestational age less than 37 weeks
* patients with a CCHD not requiring cardiac surgery with extra-corporeal circulation in the first 2 months of life
* patients with a chromosomal abnormality or genetic syndrome proven associated with CCHD

Ages: 0 Months to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Measurement of the association between age at surgery (days of life) and scores (mean = 100, standard deviation = 15) obtained on the Bayley II test | 12 months
  Measurement of the association between age at surgery (days of life) and scores (mean = 100, standard deviation = 15) obtained on the Bayley II test for each subtest: motor, cognitive and language. This association will be evaluated by a correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice DESNOUS, MD, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No